CLINICAL TRIAL: NCT05824091
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Trial in Healthy Adults to Evaluate the Safety, Tolerability, and PK of MK-7762
Brief Title: Safety, Tolerability, Pharmacokinetics (PK), and Food Effect of MK-7762 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gates MRI-TBD09-101
Record Dates: First submitted 2023-03-22; First posted 2023-04-21 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-7762 (TBD09) (Experimental): In Part 1 of the trial (SAD/FE), up to five sequential cohorts will be enrolled to evaluate up to five escalating single doses of MK-7762; 8 participants in each cohort will be randomized (3:1) to receive MK-7762 or placebo. A sixth cohort will evaluate the effect of food on PK of single doses of MK-7762 utilizing an open-label, two-period design in 8 participants.
  Interventions: Drug: MK-7762 (TBD09)
- Placebo (Placebo Comparator): Participants will receive placebos matched to MK-7762 (TBD09).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: MK-7762 (TBD09) — Cohort 1: 50 mg Cohort 2: 150 mg Cohort 3: 300 mg Cohort 4: 600 mg Cohort 5: TBD Cohort 6: TBD
  Arms: MK-7762 (TBD09)
Other: Placebo — A subset of participants from each of the 6 dosing cohorts will receive placebo.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, and pharmacokinetics of single and then multiple doses of MK-7762 (TBD09) in healthy volunteers in the context of a first-in-human study. The effect of food on the rate and extent of absorption of a single oral dose of MK-7762 (TBD09) will also be evaluated.

DETAILED DESCRIPTION:
This is a 2-part blinded, placebo-controlled, combined single ascending dose with a food effect cohort and multiple ascending dose trial to be conducted in one trial center in the United States.

Part 1 has a single ascending dose (SAD) design with up to 5 planned dose levels. Based on the interim PK results reviewed for the dose escalation decisions, a dose will be selected for administration to a sixth cohort both in fed and fasted states to evaluate the effect of food on MK-7762 (TBD09).

Safety will be assessed throughout the study; cardiac monitoring/serial ECGs and serial blood samples will be collected for the safety and PK assessment of MK7762 (TBD09). Dose escalation to the next cohort (i.e., dose level) will not take place until the Sponsor, in conjunction with the Principal Investigator, has determined that adequate safety, tolerability (and PK for the later cohorts) from the previous cohort has been demonstrated to permit proceeding to the next cohort.

Interim PK analyses will be performed for the dose escalation decisions (after cohorts 1 and 2 are completed), to select the intermediate dose for the food effect cohort, and to reconsider the sampling time points as the trial progresses. All samples will be sent for analysis and the bioanalytical lab will be unblinded and only run the analysis on active treatment participants. At the escalation meetings, PK analyses from active treatment participants and blinded (pooled) safety summaries will be reviewed.

All participants in Part 1 will remain at the trial site from Day -1 until their end of-trial visit (approximately 8 days for Cohorts 1-5 and 16 days for Cohort 6).

At the end of Part 1, pharmacokinetic and unblinded safety data along with dose rationale for Part 2 will be sent to the Food and Drug Administration (FDA) for review and approval. The trial will not proceed to Part 2 until the FDA provides approval.

Part 2 has a multiple ascending dose (MAD) design. The dose cohorts for Part 2 will be determined based on model predictions to determine the steady-state Cmax exposure, and safety from Part 1.

In this MAD part, each participant will be administered MK7762 or matching placebo for 28 days with corresponding PK measurements. Three dose cohorts are planned. After each dose cohort, the Sponsor and Investigator will review the PK and safety data before proceeding to the next dose level.

ELIGIBILITY:
Inclusion Criteria:

To be included in this trial, an individual must satisfy all the following criteria:

1. Is ≥ 19 to ≤ 55 years of age.
2. Is healthy as determined by the Investigator via medical history and clinical examination before enrollment in the trial.
3. Can understand and comply with the trial and site procedures, understand the risks involved in the trial, and provide written informed consent before the first trial-specific procedure.
4. Can complete all Screening period evaluations and stay in the clinical research facility for the duration of the inpatient periods of the trial.
5. Has BMI between 18 and 32 kg/m2, inclusive, and body weight not less than 50 kg at Screening.
6. Has resting vital signs at Screening within the following ranges: Systolic blood pressure (SBP) ≥100 mmHg Diastolic blood pressure (DBP) ≥50 mmHg Heart rate ≤100 beats per minute (bpm) Note: If vital signs are out of range, the Investigator may obtain two additional readings within the Screening period.
7. Has a 12-lead ECG consistent with normal cardiac conduction and function at Screening, including: HR between 45 and 100 bpm (inclusive); QTcF ≤450 ms for males and ≤470 ms for females; QRS interval <120 ms; PR interval <220 ms; and morphology consistent with healthy cardiac conduction.
8. Is a nonsmoker within the previous 6 months before Screening, and does not use tobacco containing, or nicotine-containing products, including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, e-cigarettes, nicotine patch, or nicotine gum.
9. Has clinical chemistry, hematology, coagulation, and complete urinalysis (fasted for at least 8 hours) results at Screening within the reference range for the testing laboratory unless the out-of-range results are deemed not clinically significant by the Investigator.
10. Has negative results for hepatitis B surface antigen (HbsAg) and hepatitis C virus antibody (HCV Ab) within 3 months prior to Day -1 or at Screening.
11. Has negative test results for HIV antibody within 3 months prior to Day -1 or at Screening.
12. Has a negative urine drug screen result at Screening and on Day -1. The presence of alcohol or marijuana in the urine is not exclusionary unless the Investigator determines that the participant's marijuana use qualifies as substance abuse (see Section 5.2, Exclusion Criteria 6).
13. If individual's assigned sex at birth is female, they must be of non-childbearing potential based on either of the following: a. Is post-menopausal defined as amenorrhea for at least 12 months in absence of any exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the laboratory-defined postmenopausal range, or, b. Reports being surgically sterilized (i.e., tubal ligation, hysterectomy, bilateral oophorectomy/salpingectomy)
14. If individual is assigned male sex at birth, is not sterilized, and is sexually active with a female partner of childbearing potential, agrees to use condoms from Day -1 through 90 days after the last dose of study drug. They must also agree to not donate sperm during the trial and for 3 months (90 days) after receiving the last dose of study drug.

Exclusion Criteria:

If an individual meets any of the following criteria, they are ineligible for this trial:

1. Has current or past history of a clinically significant cardiovascular, cerebrovascular, respiratory, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the Investigator.
2. Has history of or Screening findings of abnormalities of vision, including corrected visual acuity worse than 20/25 in either eye based on Screening assessment using Snellen chart and Rosenbaum pocket chart, or color vision impairment based on Screening assessment using Ishihara plates. Candidates with ametropia corrected to 20/25 or better do not have to be excluded.
3. Has history of or Screening findings of peripheral neuropathy, such as numbness or abnormal reflexes.
4. Has history of or current clinically relevant cardiovascular disorder, such as heart failure, coronary artery disease, uncontrolled hypertension, arrhythmia, tachyarrhythmia, prolonged QT syndrome, or presence of symptom(s) strongly suggestive of such a problem, such as exertional chest pressure/pain or unexplained syncope.
5. Had an active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers. Any history of breast cancer or melanoma will be exclusionary.
6. Has history of any drug abuse within 1 year prior to Screening or has used any hard drugs (such as cocaine, phencyclidine [PCP], natural and synthetic opiates, and amphetamine derivatives) within 1 year prior to Screening. Individuals that have taken an opioid or amphetamine medication within the previous year prior to Screening that was prescribed by a healthcare provider will not be excluded unless they are currently taking the medication at the time of Screening.
7. Has history of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces [150 mL)] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening or alcohol abuse within 1 year prior to Screening.
8. Had any surgical or medical condition or history that, in the opinion of the Investigator, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to, gastric bypass or banding surgery or gastric or duodenal ulcers.
9. Is taking any of the following prohibited medications or vaccinations: a. Any prescription or over-the-counter medication, vitamin or dietary supplement, or herbal product within 14 days prior to Day -1. b. Received any vaccination within 14 days prior to Day -1, including COVID-19 vaccination.
10. Has a contraindication to study drugs or its excipients and/or history of a clinically significant allergic or anaphylactic reaction to a medication.
11. Has participated in other trials involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before Screening for the current trial and during participation in the current trial.
12. Has a positive PCR or antigen test result for COVID-19/SARS-CoV-2 at check-in to the Clinical Trials Unit.
13. Has a condition that the Investigator believes would interfere with the participant's ability to provide written informed consent, comply with trial instructions, or which might confound the interpretation of the trial results or put the participant at undue risk.
14. Has donated blood within 2 months before entering the trial or planning to donate blood during the trial or within 12 weeks after the final visit.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Safety: To characterize safety and tolerability of MK-7762 (TBD09) after administration of single doses or multiple doses in healthy adult participants. | Part 1, Cohorts 1 through 5: Day 1 through Day 7.
  Assessed by the proportion of treated participants reporting treatment-emergent adverse events (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs), assessed overall, by severity, by relationship to study drug, and by system organ class and preferred term.
Safety: To characterize safety and tolerability of MK-7762 (TBD09) after administration of single doses or multiple doses in healthy adult participants. | Part 1, Cohort 6 (Food Effect): Day 1 through last day of washout period for first dosing period; Day 1 of second dosing period through Day 7 of second dosing period.
  Assessed by the proportion of treated participants reporting treatment-emergent adverse events (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs), assessed overall, by severity, by relationship to study drug, and by system organ class and preferred term.
Safety: To characterize safety and tolerability of MK-7762 (TBD09) after administration of single doses or multiple doses in healthy adult participants. | Part 2, Cohorts 1-3: Day 1 through Day 33.
  Assessed by the proportion of treated participants reporting treatment-emergent adverse events (TEAEs), serious AEs (SAEs), and AEs of special interest (AESIs), assessed overall, by severity, by relationship to study drug, and by system organ class and preferred term.
Safety: To characterize laboratory results after administration of single doses or multiple doses of MK-7762 (TBD09). | Part 1
  In treated participants, summaries (descriptive statistics and frequencies) of safety laboratory measures (by visit, worst grade, grade shift from baseline) according to the same windows defined above for AEs.
Safety: To characterize laboratory results after administration of single doses or multiple doses of MK-7762 (TBD09). | Part 2
  In treated participants, summaries (descriptive statistics and frequencies) of safety laboratory measures (by visit, worst grade, grade shift from baseline) according to the same windows defined above for AEs.
Safety: To characterize electrocardiogram (ECG) parameters after administration of single doses or multiple doses of MK-7762 (TBD09). | Part 1
  In treated participants, 12-lead ECG parameters including ECG QT interval with correction factors, heart rate, RR interval, PR interval (by visit, change from baseline) according to the same windows defined above for AEs.
Safety: To characterize electrocardiogram (ECG) parameters after administration of single doses or multiple doses of MK-7762 (TBD09). | Part 2
  In treated participants, 12-lead ECG parameters including ECG QT interval with correction factors, heart rate, RR interval, PR interval (by visit, change from baseline) according to the same windows defined above for AEs.
Safety: To characterize vital signs after administration of single doses or multiple doses of MK-7762 (TBD09). | Part 1
  In treated participants, vital signs (by visit, change from baseline) according to the same windows defined above for AEs.
Safety: To characterize vital signs after administration of single doses or multiple doses of MK-7762 (TBD09). | Part 2
  In treated participants, vital signs (by visit, change from baseline) according to the same windows defined above for AEs.

SECONDARY OUTCOMES:
Oral Pharmacokinetics (PK) of MK-7762 (TBD09) following a single dose and multiple doses | Day 1, Day 28
  Maximum plasma drug concentration (Cmax)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Day 1, Day 28
  Time to maximum plasma drug concentration (Tmax)
Oral PK of MK-7762 (TBD09) following single dose | Part 1 Day 1
  Area under the concentration-time curve (AUC) calculated over the first 24h (AUC(0-24)
Oral PK of MK-7762 (TBD09) following multiple doses | Part 2 Day 28
  AUC calculated over a dosing interval (AUCTau)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 1 Day 1
  AUC calculated to last quantifiable observed sample (AUC(0-last))
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 2 Day 28
  AUC calculated to last quantifiable observed sample (AUC(0-last))
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 1 Day 1
  AUC extrapolated to infinity (AUC(0-inf))
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 2 Day 28
  AUC extrapolated to infinity (AUC(0-inf))
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 1 Day 1
  Terminal elimination half-life (t½)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 2 Day 28
  Terminal elimination half-life (t½)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 1 Day 1
  Oral clearance (CL/F)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 2 Day 28
  Oral clearance (CL/F)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 1 Day 1
  Oral volume of distribution (Vd/F)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 2 Day 28
  Oral volume of distribution (Vd/F)
Oral PK of MK-7762 (TBD09) following a single dose and multiple doses | Part 2 Day 1, Day 28
  Accumulation ratio (AUCTau / AUC(0-24))
Oral PK of MK-7762 (TBD09) following a single dose in a fasted state and fed state | Part 1, Cohort 6, Day 1
  AUC(0-inf) fasted state / AUC(0-inf) fed state
Oral PK of MK-7762 (TBD09) following a single dose in a fasted state and fed state | Part 1, Cohort 6, Day 1
  Cmax fasted state / Cmax fed state

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates MRI
Locations (1):
- Investigational Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes